CLINICAL TRIAL: NCT01719419
Title: The Effect of Modified Sham Feeding With Orlistat in Overweight and Obese Subjects: A Pilot Study
Brief Title: The Effect of Modified Sham Feeding With Orlistat in Overweight and Obese Subjects
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Frank Greenway, Principal Investigaator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PBRC 12014
Record Dates: First submitted 2012-10-30; First posted 2012-11-01 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight | interventions — Orlistat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Experimental): Fatty food intake on the day the Modified sham feeding technique with placebo compared to the day modified sham feeding with orlistat.
  Interventions: Drug: Placebo
- Orlistat (Experimental): Fatty food intake on the day of the modified sham feeding technique with orlistat compared to the day with placebo.
  Interventions: Drug: Orlistat

INTERVENTIONS:
Drug: Placebo — Measured fatty food intake and appetite at a single lunch meal after the administration of modified sham feeding technique with placebo.
  Arms: Placebo
Drug: Orlistat — Measured fatty food intake and appetite at a single lunch meal after the administration of modified sham feeding technique with orlistat.
  Arms: Orlistat

SUMMARY:
The purpose of this study is to determine if the drug orlistat (Alli, Xenical) decreases the taste for fat in humans.

DETAILED DESCRIPTION:
One screening visit and Testing Visits 1 and 2: Approximately 1-2 hours (Fasting - You will have nothing to eat or drink (except water or medications) after midnight before the test visit.) If you qualify for the study, you will return to Pennington Biomedical Research Center for the test visit

* You will be given a questionnaire to screen for allergies or cold symptoms.
* Women will answer a questionnaire based on their menstrual cycle.
* Before eating, you will be given instructions on how to use the study medication. You will swish about 2 teaspoons of a solution in your mouth for 30 seconds and then spit it out (like mouthwash).
* Just before eating, you will be given another brief questionnaire judging your appetite.
* You will be given the test meal. You will be allowed to eat as much or as little as you like during a 20-minute eating period.
* 30 minutes after starting your meal you will be given the brief questionnaire again to judge your appetite.
* You will return in 1 month to complete test visit 2.

ELIGIBILITY:
Inclusion Criteria:

* Are a healthy male or female,
* Are between 18 to 70 years of age,
* Have a body mass index between 25-35 kg/m2

Exclusion Criteria:

* Are a female who is pregnant or nursing,
* Are a restrained eater (determined using a questionnaire),
* Have any current illnesses such as an infection,
* Have any serious medical problems including kidney, liver, heart or lung disease,

  * Use medications known to increase appetite,
  * Are taking any medication that has not been on the same dose for at least 30 days,
  * Dislike the test food.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Does orlistat decreases the taste for fatty food intake | 1 month
  * Before eating, you will be given instructions on how to use the study medication. You will swish about 2 teaspoons of a solution in your mouth for 30 seconds and then spit it out (like mouthwash).
  * Just before eating, you will be given another brief questionnaire judging your appetite.
  * You will be given the test meal. You will be allowed to eat as much or as little as you like during a 20-minute eating period.
  * 30 minutes after starting your meal you will be given the brief questionnaire again to judge your appetite.
  * You will return in 1 month to complete test visit 2.

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States